CLINICAL TRIAL: NCT06763406
Title: The Effects of Schroth Based Exercise Therapy in Adolescents with Pectus Excavatum
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Busra Kandemir, Principal Investigator, Hacettepe University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KA-22069/ 11.04.2023
Record Dates: First submitted 2024-12-04; First posted 2025-01-08 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Pectus Excavatum; Pectus Excavatum Deformity; Funnel Chest; Chest Deformities
Keywords: Funnel chest; Pectus excavatum; Exercise; Exercise therapy; Vacuum; Tissue expansion devices
MeSH Terms: conditions — Funnel Chest; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- vacuum only (No Intervention)
- Vacuum plus exercise (Experimental)
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Due to the limited research on exercise approaches for pectus excavatum, further investigation in this field is needed. This study aims to explore the impact of Schroth-based exercise therapy on adolescents with pectus excavatum.
  Arms: Vacuum plus exercise

SUMMARY:
Research on exercise methods for pectus excavatum (PE) is limited, highlighting the need for further studies. This study investigated the effects of Schroth-based exercise therapy combined with vacuum treatment in 35 adolescents with PE, divided into a vacuum + exercise group (n=19) and a vacuum-only group (n=16). Outcomes included deformity severity, sagittal posture, thoracic cage and spinal mobility, muscle endurance, and quality of life. The combination therapy significantly improved sagittal spinal posture (craniovertebral, thoracic, thoracolumbar, lumbar angles) and deformity-specific quality of life (Nuss Questionnaire scores) compared to vacuum-only treatment.

ELIGIBILITY:
Inclusion Criteria:

* having pectus excavatum
* being 10-18 years
* having Haller index more than 2.5

Exclusion Criteria:

* Individuals with pectus excavatum associated with a syndrome Individuals with mixed deformity
* Individuals who have previously received any conservative treatment or surgery for chest deformity or spinal issues
* Individuals with neuromuscular, rheumatic, or chronic systemic diseases

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 35 (Actual)
Dates: Start 2023-04-15 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Primary Outcome Measure 1: Deformity Severity | 12 weeks
  Primary Outcome Measure 1: Deformity Severity Measurement: Anthropometric Index (cm) Details: Repeated, in cm. Time frame: The assessment will be conducted during the first week of treatment and 12 weeks after treatment
Primary Outcome Measure 2: Sagittal Spinal Posture | 12 weeks
  Primary Outcome Measure 2: Sagittal Spinal Posture Measurement: Lateral Photos (°) Details: In degrees Time Frame:The assessment will be conducted during the first week of treatment and 12 weeks after treatment
Primary Outcome Measure 3: Disease-Specific QoL | 12 weeks
  Primary Outcome Measure 3: Disease-Specific QoL Measurement: Nuss Questionnaire (1-4) Details: Higher = better Time Frame: The assessment will be conducted during the first week of treatment and 12 weeks after treatment
Primary Outcome Measure 4: General QoL | 12 weeks
  Primary Outcome Measure 4: General QoL Measurement: PedsQL (0-100) Details: Higher = better Time Frame: The assessment will be conducted during the first week of treatment and 12 weeks after treatment

SECONDARY OUTCOMES:
Secondary Outcome Measure 1: Thoracic Cage Mobility | 12 weeks
  Secondary Outcome Measure 1: Thoracic Cage Mobility Measurement: Chest Circumference (cm) Details: In cm Time Frame: The assessment will be conducted during the first week of treatment and 12 weeks after treatment
Secondary Outcome Measure 2: Spinal Mobility | 12 weeks
  Secondary Outcome Measure 2: Spinal Mobility Measurement: Sit-and-Reach (cm) Details: Highest value Time Frame: The assessment will be conducted during the first week of treatment and 12 weeks after treatment
Secondary Outcome Measure 3: Lumbar Mobility | 12 weeks
  Secondary Outcome Measure 3: Lumbar Mobility - Measurement: Modified Schober (cm) Details: Difference in cm Time Frame: The assessment will be conducted during the first week of treatment and 12 weeks after treatment
Secondary Outcome Measure 4: Muscle Endurance (Sit-Ups) | 12 weeks
  Secondary Outcome Measure 4: Muscle Endurance (Sit-Ups) Measurement: Sit-Up (reps/30s) Details: Repetitions Time Frame: The assessment will be conducted during the first week of treatment and 12 weeks after treatment
Secondary Outcome Measure 5: Muscle Endurance (Lateral Bridge) | 12 weeks
  Secondary Outcome Measure 5: Muscle Endurance (Lateral Bridge) Measurement: Lateral Bridge (s) Details: Duration Time Frame: The assessment will be conducted during the first week of treatment and 12 weeks after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe Uuniversity, Ankara, altındağ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No